CLINICAL TRIAL: NCT04091646
Title: A Phase 2b, 8-Week, Parallel Group, Double Blind, Vehicle-Controlled Study of the Safety and Efficacy of ARQ-154 Foam 0.3% Administered QD in Subjects With Seborrheic Dermatitis
Brief Title: Safety and Efficacy of ARQ-154 Foam in Subjects With Seborrheic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arcutis Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARQ-154-203
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Results first posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Seborrheic Dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Roflumilast Foam 0.3% (Active Comparator): Participants apply roflumilast foam 0.3% once daily (QD) to all areas of seborrheic dermatitis once daily for 8 weeks.
  Interventions: Drug: Roflumilast Foam 0.3%
- Vehicle Foam (Placebo Comparator): Participants apply inactive vehicle foam matched to roflumilast foam QD for 8 weeks.
  Interventions: Drug: Vehicle foam

INTERVENTIONS:
Drug: Roflumilast Foam 0.3% — Roflumilast foam for topical application.
  Other Names: ARQ-154
  Arms: Roflumilast Foam 0.3%
Drug: Vehicle foam — Vehicle foam for topical application.
  Other Names: Placebo
  Arms: Vehicle Foam

SUMMARY:
This was a parallel group, double blind, vehicle-controlled study assessed the safety and efficacy of roflumilast foam (ARQ-154) vs placebo foam in participants with seborrheic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Participants legally competent to sign and give informed consent.
2. Males and females ages 18 years and older (inclusive) at the time of consent.
3. Clinical diagnosis of seborrheic dermatitis of at least 3 months duration as determined by the Investigator. Stable disease for the past 4 weeks.
4. Seborrheic dermatitis of the scalp and/or face and/or trunk and/or intertriginous areas.
5. An Investigator Global Assessment (IGA) of disease severity of at least Moderate ('3') at Baseline.
6. Overall Assessment of Erythema and Overall Assessment of Scaling scores of at least Moderate ('2') at Baseline.
7. Females of childbearing potential (FOCBP) must have a negative serum pregnancy test at Screening (Visit 1) and a negative urine pregnancy test at Baseline (Visit 2).
8. Females of non-childbearing potential must either be post-menopausal with spontaneous amenorrhea for at least 12 months or have undergone surgical sterilization.
9. Subjects in good health as judged by the Investigator, based on medical history, physical examination, vital signs, serum chemistry labs, hematology values, and urinalysis.
10. Subjects are considered reliable and capable of adhering to the Protocol and visit schedule according to the Investigator judgment.

Exclusion Criteria:

1. Subjects who cannot discontinue treatment with therapies for the treatment of seborrheic dermatitis prior to the Baseline visit and during the study according to Excluded Medications and Treatments.
2. Planned excessive exposure of treated area(s) to either natural or artificial sunlight, tanning bed or other LED.
3. Subjects who cannot discontinue the use of strong P-450 cytochrome inhibitors e.g., indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, nefazodone, saquinavir, suboxone and telithromycin for two weeks prior to the Baseline visit (Visit 2) and during the study.
4. Subjects who cannot discontinue the use of strong P-450 cytochrome inducers e.g., efavirenz, nevirapine, glucocorticoids, barbiturates (including phenobarbital), phenytoin, rifampin, and carbamazepine for two weeks prior to the Baseline visit (Visit 2) and during the study.
5. Subjects with PHQ-8 ≥10 at Screening or Baseline visits.
6. Previous treatment with ARQ-151 and ARQ-154.
7. Subjects who have received oral roflumilast (Daliresp®, Daxas®) or other PDE-4 inhibitors (apremilast) within the past 4 weeks.
8. Known allergies to excipients in ARQ-154 foam.
9. Known or suspected: severe renal insufficiency or moderate to severe hepatic disorders; hypersensitivity to component(s) of the investigational products; or history of severe depression, suicidal ideation, or Baseline/Screening C-SSRS indicative of suicidal ideation, whether lifetime or recent/current.
10. Subjects with a history of a major surgery within 8 weeks prior to Baseline (Visit 2) or has a major surgery planned during the study.
11. Subjects with any condition on the treatment area which, in the opinion of the Investigator, could confound efficacy measurements.
12. Subjects unable to apply product to the scalp due to physical limitations.
13. Females who are pregnant, wishing to become pregnant during the study, or are breast-feeding.
14. A clinically relevant history of abuse of alcohol or other drugs, at the discretion of the Investigator.
15. Subjects who are unable to communicate, read or understand the local language, or who display another condition, which in the Investigator's opinion, makes them unsuitable for clinical study participation.
16. Subjects who are family members of the clinical study site, clinical study staff, or sponsor, or family members of enrolled subjects.
17. Any condition that in the Investigator's assessment would preclude the subject from participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Berk, MD, Study Director — Arcutis Biotherapeutics, Inc.
Locations (24):
- United States (22):
  - Arcutis Biotherapeutics Clinical Site 19, Fremont, California
  - Arcutis Biotherapeutics Clinical Site 21, Santa Monica, California
  - Arcutis Biotherapeutics Clinical Site 42, Coral Gables, Florida
  - Arcutis Biotherapeutics Clinical Site 24, Miami, Florida
  - Arcutis Biotherapeutics Clinical Site 12, Tampa, Florida
  - Arcutis Biotherapeutics Clinical Site 10, Rolling Meadows, Illinois
  - Arcutis Biotherapeutics Clinical Site 22, Plainfield, Indiana
  - Arcutis Biotherapeutics Clinical Site 15, Louisville, Kentucky
  - Arcutis Biotherapeutics Clinical Site 28, Rockville, Maryland
  - Arcutis Biotherapeutics Clinical Site 40, Clinton Township, Michigan
  - Arcutis Biotherapeutics Clinical Site 20, Detroit, Michigan
  - Arcutis Biotherapeutics Clinical Site 14, Fridley, Minnesota
  - Arcutis Biotherapeutics Clinical Site 23, High Point, North Carolina
  - Arcutis Biotherapeutics Clinical Site 18, Bexley, Ohio
  - Arcutis Biotherapeutics Clinical Site 29, Portland, Oregon
  - Arcutis Biotherapeutics Clinical Site 27, Pittsburgh, Pennsylvania
  - Arcutis Biotherapeutics Clinical Site 13, Arlington, Texas
  - Arcutis Biotherapeutics Clinical Site 11, Austin, Texas
  - Arcutis Biotherapeutics Clinical Site 41, College Station, Texas
  - Arcutis Biotherapeutics Clinical Site 25, Houston, Texas
  - Arcutis Biotherapeutics Clinical Site 26, Pflugerville, Texas
  - Arcutis Biotherapeutics Clinical Site 17, Norfolk, Virginia
- Canada (2):
  - Arcutis Biotherapeutics Clinical Site 31, Markham, Ontario
  - Arcutis Biotherapeutics Clinical Site 30, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zirwas MJ, Draelos ZD, DuBois J, Kircik LH, Moore AY, Stein Gold L, Alonso-Llamazares J, Bukhalo M, Bruce S, Eads K, Green LJ, Guenthner ST, Ferris LK, Forman SB, Kempers SE, Lain E, Lynde CW, Pariser DM, Toth DP, Yamauchi PS, Higham RC, Krupa D, Burnett P, Berk DR. Efficacy of Roflumilast Foam, 0.3%, in Patients With Seborrheic Dermatitis: A Double-blind, Vehicle-Controlled Phase 2a Randomized Clinical Trial. JAMA Dermatol. 2023 Jun 1;159(6):613-620. doi: 10.1001/jamadermatol.2023.0846. PMID 37133856

RESULTS

PARTICIPANT FLOW:
Groups:
- Roflumilast Foam 0.3%: Participants apply roflumilast foam 0.3% once daily for 8 weeks.
- Vehicle Foam: Participants apply vehicle foam matched to roflumilast foam once daily for 8 weeks.
Period: Overall Study
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Started | 154 | 72
Completed | 141 | 67
Not Completed | 13 | 5
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 6 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Participant Incarcerated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam | Total
Number analyzed (Participants) | 154 | 72 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (17.01) | 44.2 (16.27) | 44.9 (16.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 32 | 110
  Male | 76 | 40 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 16 | 45
  Not Hispanic or Latino | 125 | 56 | 181
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American-Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 1 | 8
  Black or African-American | 17 | 6 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 123 | 62 | 185
  Other | 1 | 2 | 3
  More than One Race | 5 | 1 | 6
Investigator Global Assessment (IGA) Baseline Score [Count of Participants; unit: Participants] — The IGA is 5-point scale assessing the severity of seborrheic dermatitis, with scores ranging from 0 ('completely clear') to 4 ('severe'), with higher scores indicating greater severity.
  Participants
    0 Completely Clear | 0 | 0 | 0
    1 Almost Clear | 0 | 0 | 0
    2 Mild | 0 | 0 | 0
    3 Moderate | 141 | 69 | 210
    4 Severe | 13 | 3 | 16
Worst Itch Numerical Rating Scale (WI-NRS) Baseline Score [Count of Participants; unit: Participants] — The WI-NRS is a simple, single-item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the subject experienced in the previous 24 hours. Higher scores indicate greater severity.
  Participants
    0 | 7 | 2 | 9
    1 | 6 | 2 | 8
    2 | 9 | 5 | 14
    3 | 7 | 4 | 11
    4 | 18 | 8 | 26
    5 | 13 | 11 | 24
    6 | 20 | 5 | 25
    7 | 27 | 17 | 44
    8 | 24 | 16 | 40
    9 | 14 | 0 | 14
    10 | 9 | 2 | 11
Overall Assessment of Erythema Baseline Score [Count of Participants; unit: Participants] — The Overall Assessment of Erythema is a simple, single-item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("None: no evidence of erythema.") to 3 ("Severe: Intense (fiery red) erythema."). Higher scores indicate greater severity.
  Participants
    None | 0 | 0 | 0
    Mild | 0 | 0 | 0
    Moderate | 135 | 66 | 201
    Severe | 19 | 6 | 25
Overall Assessment of Scaling Baseline Score [Count of Participants; unit: Participants] — The Overall Assessment of Scaling is a simple, single-item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("No scaling: No scaling evident on lesions.") to 3 ("Severe: Coarse, thick scales, with flaking into clothes or skin."). Higher scores indicate greater severity.
  Participants
    None | 0 | 0 | 0
    Mild | 0 | 0 | 0
    Moderate | 130 | 58 | 188
    Severe | 24 | 14 | 38

OUTCOME MEASURES:

1. Primary Outcome: Achievement of Investigator Global Assessment (IGA) Success at Week 8
Description: The number of participants achieving "success" in IGA assessment of disease severity at Week 8 is presented for each arm. Success was defined as achievement of an IGA score of 0 ('completely clear') or 1 ('almost clear'), accompanied by a ≥2-grade improvement from baseline IGA score. The IGA is 5-point scale assessing the severity of Seborrheic Dermatitis, with scores ranging from 0 ('completely clear') to 4 ('severe'), and higher scores indicate greater severity. The IGA scores are based on observed data, whereas odds ratio and p-values were calculated using multiple imputation of missing values.
Time Frame: Week 8
Population: All randomized participants are included, with the exception of those who missed the Week 8 assessment due to COVID-19 disruption.
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 141 | 66
Participants | 104 | 27
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; IGA Success at Week 8 Odds Ratio; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Stratification by pooled study site and baseline IGA per randomization with multiple imputation of missing data; Odds Ratio (OR) = 4.95, 95% CI 2-sided [2.51 to 9.76] — Common OR stratified by pooled study site and baseline IGA per randomization with multiple imputation of missing data

2. Secondary Outcome: Achievement of IGA Success at Weeks 2 and 4
Description: The number of participants achieving "success" in IGA assessment of disease severity at Weeks 2 and 4 is presented for each arm. Success was defined as achievement of an IGA score of 0 ('completely clear') or 1 ('almost clear'), accompanied by a ≥2-grade improvement from baseline IGA score. The IGA is 5-point scale assessing the severity of Seborrheic Dermatitis, with scores ranging from 0 ('completely clear') to 4 ('severe'), and higher scores indicate greater severity. The IGA scores are based on observed data, whereas odds ratio and p-values were calculated using multiple imputation of missing values.
Time Frame: Weeks 2 and 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 151 | 68
Participants
  Week 2 | 51 | 10
  Week 4: number analyzed (Participants) | 143 | 67
  Week 4 | 81 | 19
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; IGA Success at Week 2 Odds Ratio; Test type: Superiority; p = 0.0033, Cochran-Mantel-Haenszel; Stratification by pooled study site and baseline IGA per randomization with multiple imputation of missing data; Odds Ratio (OR) = 3.31, 95% CI 2-sided [1.46 to 7.52] — Common OR stratified by pooled study site and baseline IGA per randomization with multiple imputation of missing data
Statistical Analysis 2: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; IGA Success at Week 4 Odds Ratio; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Stratification by pooled study site and baseline IGA per randomization with multiple imputation of missing data; Odds Ratio (OR) = 3.78, 95% CI 2-sided [1.94 to 7.38] — Common OR stratified by pooled study site and baseline IGA per randomization with multiple imputation of missing data

3. Secondary Outcome: Change From Baseline in Overall Assessment of Erythema Score
Description: The mean (SD) change from baseline in Overall Assessment of Erythema score at Weeks 2, 4, and 8 is shown. The Erythema Assessment is a simple, single-item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("None: no evidence of erythema.") to 3 ("Severe: Intense [fiery red] erythema."). Higher scores indicate greater severity.
Time Frame: Weeks 2, 4, and 8
Population: All randomized participants who provided data are included, with the exception of those who missed the Week 8 assessment due to COVID-19 disruption.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 151 | 68
score on a scale
  Week 2 | -1.0 (0.73) | -0.4 (0.65)
  Week 4: number analyzed (Participants) | 143 | 67
  Week 4 | -1.3 (0.73) | -0.7 (0.68)
  Week 8: number analyzed (Participants) | 141 | 66
  Week 8 | -1.4 (0.78) | -0.8 (0.85)
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Week 2 Erythema Score; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Week 4 Erythema Score; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Week 8 Erythema Score; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Achievement of Overall Assessment of Erythema Success
Description: The number of participants achieving "success" in Overall Assessment of Erythema at Weeks 2, 4, and 8 is presented for each arm. Success was defined as achievement of an overall score of 0 or 1 plus a ≥2 grade improvement from Baseline. The Overall Assessment of Erythema is a simple, single-item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("None: no evidence of erythema.") to 3 ("Severe: Intense [fiery red] erythema."). Higher scores indicate greater severity.
Time Frame: Weeks 2, 4, and 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 151 | 68
Participants
  Week 2 | 34 | 4
  Week 4: number analyzed (Participants) | 143 | 67
  Week 4 | 51 | 7
  Week 8: number analyzed (Participants) | 141 | 66
  Week 8 | 63 | 14
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Erythema Success at Week 2; Test type: Superiority; p = 0.0065, Cochran-Mantel-Haenszel; Stratification by pooled study site and baseline IGA per randomization with no imputation of missing data; Odds Ratio (OR) = 5.05, 95% CI 2-sided [1.49 to 17.13]
Statistical Analysis 2: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Erythema Success at Week 4; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel; Stratification by pooled study site and baseline IGA per randomization with no imputation of missing data; Odds Ratio (OR) = 5.36, 95% CI 2-sided [2.15 to 13.38]
Statistical Analysis 3: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Erythema Success at Week 8; Test type: Superiority; p = 0.0021, Cochran-Mantel-Haenszel; Stratification by pooled study site and baseline IGA per randomization with no imputation of missing data; Odds Ratio (OR) = 3.15, 95% CI 2-sided [1.50 to 6.63]

5. Secondary Outcome: Change From Baseline in Overall Assessment of Scaling Score
Description: The mean (SD) change from baseline in Overall Assessment of Scaling score at Weeks 2, 4, and 8 is shown. The Overall Assessment of Scaling is a simple, single-item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("No scaling: No scaling evident on lesions.") to 3 ("Severe: Coarse, thick scales, with flaking into clothes or skin."). Higher scores indicate greater severity.
Time Frame: Weeks 2, 4, and 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 151 | 68
Score on a scale
  Week 2 | -1.0 (0.77) | -0.6 (0.78)
  Week 4: number analyzed (Participants) | 143 | 67
  Week 4 | -1.3 (0.76) | -0.8 (0.81)
  Week 8: number analyzed (Participants) | 141 | 66
  Week 8 | -1.5 (0.75) | -1.0 (0.83)
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Week 2 Scaling Score; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Week 4 Scaling Score; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Week 8 Scaling Score; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Achievement of Overall Assessment of Scaling Success
Description: The number of participants achieving "success" in Overall Assessment of Scaling score at Weeks 2, 4, and 8 is presented for each arm. Success was defined as achievement of an Overall Assessment of Scaling score of 0 or 1 plus a ≥2 grade improvement from Baseline. The Overall Assessment of Scaling is a simple, single-item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("No scaling: No scaling evident on lesions.") to 3 ("Severe: Coarse, thick scales, with flaking into clothes or skin."). Higher scores indicate greater severity.
Time Frame: Weeks 2, 4, and 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 151 | 68
Participants
  Week 2 | 40 | 10
  Week 4: number analyzed (Participants) | 143 | 67
  Week 4 | 59 | 14
  Week 8: number analyzed (Participants) | 141 | 66
  Week 8 | 63 | 14
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Scaling Success at Week 2; Test type: Superiority; p = 0.0759, Cochran-Mantel-Haenszel; Stratification by pooled study site and baseline IGA per randomization with no imputation of missing data; Odds Ratio (OR) = 1.98, 95% CI 2-sided [0.90 to 4.33] — Common OR stratified by pooled study site and baseline IGA per randomization with no imputation of missing data
Statistical Analysis 2: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Scaling Success at Week 4; Test type: Superiority; p = 0.0122, Cochran-Mantel-Haenszel; Stratification by pooled study site and baseline IGA per randomization with no imputation of missing data; Odds Ratio (OR) = 2.33, 95% CI 2-sided [1.18 to 4.61] — Common OR stratified by pooled study site and baseline IGA per randomization with no imputation of missing data
Statistical Analysis 3: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; Scaling Success at Week 8; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Stratification by pooled study site and baseline IGA per randomization with no imputation of missing data; Odds Ratio (OR) = 3.37, 95% CI 2-sided [1.74 to 6.55] — Common OR stratified by pooled study site and baseline IGA per randomization with no imputation of missing data

7. Secondary Outcome: Change From Baseline in Worst Itch Numeric Rating Scale (WI-NRS) Score
Description: The change from baseline in WI-NRS is shown. The WI-NRS is a simple, single-item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the subject experienced in the previous 24 hours. Negative values represent a decrease in worst itch from baseline, and positive values indicate an increase.
Time Frame: Weeks 2, 4, and 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 151 | 67
score on a scale
  Week 2 | -3.0 (2.80) | -1.7 (2.08)
  Week 4: number analyzed (Participants) | 148 | 66
  Week 4 | -3.5 (2.72) | -1.9 (2.22)
  Week 8: number analyzed (Participants) | 141 | 66
  Week 8 | -3.7 (2.83) | -2.0 (2.37)

8. Secondary Outcome: Achievement of WI-NRS Success
Description: The number of participants achieving WI-NRS "success" at Weeks 2, 4, and 8 is presented. Success was defined as achievement of a ≥4-point improvement from baseline WI-NRS score. The WI-NRS is a simple, single-item scale to assess the subject-reported severity of this symptom, on a scale ranging from 0 ("no itch") to 10 ("worst imaginable itch") the subject experienced in the previous 24 hours.
Time Frame: Weeks 2, 4, and 8
Population: All randomized participants who provided data are included, with the exception of those who missed the Week 8 assessment due to COVID-19 disruption or those with baseline WI-NRS <4.
Measure: Count of Participants; unit: Participants
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
Number analyzed (Participants) | 123 | 56
Participants
  Week 2 | 65 | 13
  Week 4: number analyzed (Participants) | 120 | 53
  Week 4 | 70 | 15
  Week 8: number analyzed (Participants) | 113 | 53
  Week 8 | 73 | 18
Statistical Analysis 1: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; WI-NRS Success at Week 2; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel; Stratification by pooled study site and baseline IGA per randomization with no imputation of missing data; Odds Ratio (OR) = 3.62, 95% CI 2-sided [1.72 to 7.63] — Common OR stratified by pooled study site and baseline IGA per randomization with no imputation of missing data
Statistical Analysis 2: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; WI-NRS Success at Week 4; Test type: Superiority; p = 0.0009, Cochran-Mantel-Haenszel; Stratification by pooled study site and baseline IGA per randomization with no imputation of missing data; Odds Ratio (OR) = 3.30, 95% CI 2-sided [1.63 to 6.68] — Common OR stratified by pooled study site and baseline IGA per randomization with no imputation of missing data
Statistical Analysis 3: Comparison: Roflumilast Foam 0.3% vs Vehicle Foam; WI-NRS Success at Week 8; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel; Stratification by pooled study site and baseline IGA per randomization with no imputation of missing data; Odds Ratio (OR) = 3.19, 95% CI 2-sided [1.60 to 6.35] — Common OR stratified by pooled study site and baseline IGA per randomization with no imputation of missing data

ADVERSE EVENTS:
Time Frame: Up to ~63 days
Description: All participants who received ≥1 dose of study treatment are included.
Arm/Group | Roflumilast Foam 0.3% | Vehicle Foam
All-Cause Mortality (participants affected / at risk) | 0/154 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/154 | 0/72
Other Adverse Events (participants affected / at risk) | 0/154 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor is supportive of publishing clinical trial findings. The process of coordinating publication efforts is detailed in the Clinical Trial Agreement.

DOCUMENTS (2):
  • Study Protocol (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT04091646/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT04091646/SAP_001.pdf